CLINICAL TRIAL: NCT06233175
Title: Combined Open And Closed Kinetic Chain Exercises On Static And Dynamic Strength Of Hamstring And Quadriceps In Knee Osteoarthritis Patients
Brief Title: Combined Kinetic Chain Exercises on Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hadeer Ali El sayaad, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004731
Record Dates: First submitted 2024-01-20; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: static knee strength,; dynamic knee strength; combined kinetic chain exercises; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: I will assess the patient before and after end of intervention programme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator): patients take conventional trans cutaneous electrical stimulation (tens) with a frequency of 100 Hz , a pulse duration of 60 micro seconds for 20 min. ,hot backs for 15 min,stretching exercises for hamstring ,quadriceps ,calf muscles
  Interventions: Other: conventional
- interventional group (Experimental): patients take conventional tens with a frequency of 100 Hz , a pulse duration of 60 micro seconds for 20 min. ,hot backs for 15 min,stretching exercises for hamstring ,quadriceps ,calf muscles with combined kinetic chain exercises (terminal knee extension,semi squat (wall slide) ,foreword step up and down ,straight leg raise ,seated knee extension )
  Interventions: Other: combined kinetic chain exercises

INTERVENTIONS:
Other: combined kinetic chain exercises — combined kinetic chain exercises in form of wall slide ,terminal knee extension ,forward step up and down ,side step up and down ,straight leg raise ,seated knee extension ,stretching exercises , hot back and trans cutaneous electrical stimulation,
  Other Names: experimental
  Arms: interventional group
Other: conventional — stretching exercises and hot back and trans cutaneous electrical stimulation,with out combined kinetic chain exercises
  Other Names: control
  Arms: conventional group

SUMMARY:
study will be conducted at faculty of physical therapy cairo university to investigate the effect of combined kinetic chain exercises on static and dynamic hamstring and quadriceps strength in knee osteoarthritis patients

DETAILED DESCRIPTION:
the study will be conducted at faculty of physical therapy cairo university to investigate the effect of combined kinetic chain exercises on static and dynamic hamstring and quadriceps strength ,knee pain ,function ,H/Q ratio in knee osteoarthritis patients .using lafayette hand held dynamometer to measuring static strength of hamstring and quadriceps ,and free weight by Brzycki formula for measuring dynamic hamstring and quadriceps strength by determining 1 repetition maximum ,and pain measured by visual analogue scale (VAS) rating from (0 = no pain ) to (10= worst pain ) ,and function by Western Ontario and McMaster Universities Osteoarthritis Index questionnaire lower score indicate patient get better ,number of patients will be 34 divided into 2 groups ,each group will include 17 patient ,with 2 drop out according to sample size calculation ,each group will receive conventional tens for 20 min. and hot back for 15 min. and stretching exercises for hamstring,quadriceps,calf muscles ,while the experimental group will be increased by combined kinetic chain exercises

ELIGIBILITY:
Inclusion Criteria:

* the patients age from38 to 65
* recent radiographs confirming grade 2 and 3 (mild to moderate ) osteoarthritis
* primary and secondary Osteoarthritis
* both gender
* unilateral knee osteoarthritis
* pain in the knee for most days of prior month
* morning stiffness less than 30 min. in duration
* patient body mass index (BMI) between 18.5 and 29.9 kg/m2

Exclusion Criteria:

* neurological disorders
* wheelchair bound
* significant cognitive impairment
* present systemic inflammatory arthritis
* history of hip and knee arthroplasty

  * history of trauma or surgical arthroscopy of either knee in the last 6 months
* received knee intra-articular injection within the last 3 months
* under anticoagulant therapy ,recent or imminent surgery (within 3 months)

Ages: 38 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
static quadriceps strength | Evaluation will be performed prior to the first treatment session ;as a baseline measure,and at last treatment session (after 4 weeks) as a post -treatment measure
  measuring static quadriceps from sitting position at angle 60 and 90
static hamstring strength | Evaluation will be performed prior to the first treatment session ;as a baseline measure,and at last treatment session (after 4 weeks) as a post -treatment measure
  measuring static hamstring strength from sitting position at angle 60 and 90
dynamic quadriceps strength | Evaluation will be performed prior to the first treatment session ;as a baseline measure,and at last treatment session (after 4 weeks) as a post -treatment measure
  measuring dynamic quadriceps strength from sitting position by randomised free weight and Brzycki formula
dynamic hamstring strength | Evaluation will be performed prior to the first treatment session ;as a baseline measure,and at last treatment session (after 4 weeks) as a post -treatment measure
  measuring dynamic hamstring strength from prone position by randomised free weight and Brzycki formula
Hamstring /Quadriceps ((H/Q) ratio | Evaluation will be performed prior to the first treatment session ;as a baseline measure,and at last treatment session (after 4 weeks) as a post -treatment measure
  dividing static hamstring on static quadriceps strength and dynamic hamstring on dynamic quadriceps strength

SECONDARY OUTCOMES:
change in neck pain | Evaluation will be performed prior to the first treatment session ;as a baseline measure,and at last treatment session (after 4 weeks) as a post -treatment measure
  by Visual Analog Scale (VAS) , (0=no pain ) and (10=worst pain)
function | Evaluation will be performed prior to the first treatment session ;as a baseline measure,and at last treatment session (after 4 weeks) as a post -treatment measure
  BYWestern Ontario and McMaster Universities Osteoarthritis Index questionnaire ,Lower score indicate patient gets better

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt